CLINICAL TRIAL: NCT05194280
Title: Robot-assisted Donornephrectomy: Initial Results and Comparison With the Hand-assisted Laparoscopic Technique: A Retrospective Study
Brief Title: Comparison of Robot-assisted Donornephrectomy vs Hand-assisted Laparoscopic Donornephrectomy
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Dr. Mirza Idu, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: 2021_01
Record Dates: First submitted 2021-12-18; First posted 2022-01-18 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Kidney Donation; Robotic Surgery
Keywords: Donornephrectomy; Robotic-asisted donornephrectomy; hand-assisted laparoscopic donornephrectomy
MeSH Terms: interventions — Robotic Surgical Procedures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Robotic-assisted group: Group of patients that underwent a robotic-assisted donornephrectomy
  Interventions: Procedure: Robotic surgery
- Hand-assisted laparoscopic group: Group of patients that underwent a hand-assisted laparoscopic donornephrectomy.

INTERVENTIONS:
Procedure: Robotic surgery — Robotic-assisted donornephrectomy
  Groups: Robotic-assisted group

SUMMARY:
The aim of this retrospective study was to analyze donor and recipient outcomes after robotic-assisted donor nephrectomy and hand-assisted laparoscopic donornephrectomy.

DETAILED DESCRIPTION:
Living donor kidney transplantation is superior to cadaveric kidney transplantation because of the better patient and graft survival rates, better cost-effectiveness and improved quality of life of the recipient. According to the current guidelines, the laparoscopic technique of donor nephrectomy is now recommended as "the preferential technique". The advantages of the hand-assisted laparoscopic donor nephrectomy (HALDN) as compared with the conventional laparoscopy include tactile feedback, less kidney traction, rapid kidney removal and a shorter warm ischemic period. HALDN is nowadays the most frequently used technique in the U.S. for living donor nephrectomy. The laparoscopic techniques may have helped to increase the expansion of the donor pool. However, laparoscopic surgery have some disadvantages especially ergonomic inconveniences for the surgeon, which may result in decreased surgeons' performance and musculoskeletal disorders. Surgical robotics can play a role in extending surgical careers, by allowing surgeons to perform high volume laparoscopic surgery in a more ergonomic way. Robotic assistance in living donor nephrectomy can offer improved safety by enhanced control, accuracy, stability, and vision. The aim of this retrospective study was to compare the robotic assisted donor nephrectomy (RADN) with the HALDN technique with respect to donor and recipient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adult, healthy condition

Exclusion Criteria:

* Children, not suitable for kidney donation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kidney donors
Sampling Method: Non-Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-10-20 (Actual)

PRIMARY OUTCOMES:
Post-operative pain score | 0-3 days
  Visual Analogue Scale was used to measure the postoperative pain. From the operation date till discharge from the hospital

SECONDARY OUTCOMES:
Operating time | 30-300 min
  Operating time in minutes

CONTACTS AND LOCATIONS:
Overall Officials: Mirza Idu, MD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Amsterdam UMC, location AMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No